CLINICAL TRIAL: NCT02538640
Title: Determination of the Postprandial Responses to Two Cereal Foods Differing by Their SDS Content and GI Consumed Alone.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: KBE040
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Metabolism and Nutrition Disorders
Keywords: Nutrition, glycemic response, cereal products
MeSH Terms: conditions — Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-SDS biscuit (Experimental): 50 g of moist biscuit with high-SDS content and low GI with a glass of water
  Interventions: Other: High-SDS biscuit
- Low-SDS breakfast cereals (Active Comparator): 42 g of extruded cereals with no SDS and medium to high GI with a glass of water
  Interventions: Other: Low-SDS extruded cereals

INTERVENTIONS:
Other: High-SDS biscuit — Consumption of the high-SDS product (50g) alone with a glass of water
  Arms: High-SDS biscuit
Other: Low-SDS extruded cereals — Consumption of the low-SDS product (42g) alone with a glass of water
  Arms: Low-SDS breakfast cereals

SUMMARY:
This is a laboratory-based research study conducted in two parts. Open cross-over design. 2 test sessions per subject included in the study. It aims at determining the postprandial blood glucose and insulin responses to the ingestion of cereal product differing by their SDS content and GI in 20 healthy non-smoking voluntary subjects, aged from 18 to 45 years.

DETAILED DESCRIPTION:
This is a laboratory-based research study conducted in two parts. Open cross-over design. 2 test sessions per subject included in the study. It aims at determining the postprandial blood glucose and insulin responses to the ingestion of cereal product differing by their SDS content and GI in 20 healthy non-smoking voluntary subjects, aged from 18 to 45 years.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-45 years.
* Non-smoker.
* BMI values between 19-30 kg/m2 (bounds included). Around half of the subjects will be normal weight and the other half overweight.
* Ethnicity. Subjects should have the closest characteristics compared to the American population. Not less than 75% but not more than 90% of the subjects should be Caucasian. Not more than 10% of the subjects will be of Asian or Asian Indian descent. The remaining subjects will be from other ethnic groups except from Australian Aborigines.
* Healthy subjects with:

  * Normal glucose tolerance (fasting blood glucose < 6.0 mmol/L during the first test session and results of oral glucose tolerance test conducted within the last 30 days within recommendations (fasting blood glucose < 6.1 mmol/L, 120 minute glucose < 8.9 mmol/L))
  * Normal laboratory values for various measures of metabolic health (full blood count, gamma-GT, AST, ALT, glucose, TAGs, total cholesterol, HDL-cholesterol, LDL-cholesterol);
  * Normal systolic blood pressure (100-150 mmHg);
  * Normal diastolic blood pressure (60-90 mmHg);
  * Normal resting heart rate (50-90 beats per minutes after 3 minutes rest).
* Stable dietary habits; normal eating patterns; no history of eating disorders or strict dieting.
* Moderate level of physical activity (from basic daily activity to a high level of physical activity (regular physical activity at least 3 times per week)
* Able to fast for at least 10 hours the night before each test session
* Able to refrain from eating legumes and drinking alcohol the day before each test session.
* Subject covered by social security or covered by a similar system
* Subject not taking any treatment for anorexia, weight loss, or any form of treatment likely tointerfere with metabolism or dietary habits
* Subject having given written consent to take part in the study.

Exclusion Criteria:

* Following a restrictive diet.
* Family history of Diabetes Mellitus or obesity
* Suffering from any clinical, physical or mental illness.
* Suffering from any food allergies or hypersensitivities (wheat, milk, egg, nuts, etc).
* Taking any regular prescription medication at the time of inclusion (except regular oral contraception medication)
* Subject from the Australian Aboriginal ethnicity.
* Female who is pregnant (positive test results), lactating, planning pregnancy or not using acceptable contraceptive.
* Females who consistently suffer from premenstrual tension and marked changes in appetite during their menstrual cycle.
* Subject having taken part in another clinical trial within the last week.
* Subject currently taking part in another clinical trial or being in the exclusion period of another clinical trial.
* Subject undergoing general anaesthesia in the month prior to inclusion.
* Subject in a situation which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Glycemic Response over 2 hours | 2 hours
  iAUC of glycemia over 2 first hours of postprandial period

SECONDARY OUTCOMES:
Glycemic response | 4 hours
  Postprandial changes in glycaemia over 3 hours (iAUC [0-180]), 4h (iAUC[0-240]), during the second part of the morning (iAUC [120-240] and iAUC[180-240]) following the intake of the test products will be analysed
Blood glucose kinetic | 4 hours
  Postprandial kinetic of glycemia over the full postprandial period (analysis time by time)
Insulinemic response | 4 hours
  Postprandial changes in insulinemia over 2 hours (iAUC [0-120]), 3 hours (iAUC [0-180]), 4h (iAUC[0-240]), during the second part of the morning (iAUC [120-240] and iAUC [180-240]) following the intake of the test products will be analysed.
Blood insulin kinetic | 4 hours
  Postprandial kinetic of insulinemia over the full postprandial period (analysis time by time)
Blood glucose peak | 4 hours
  Maximal concentration and delta between maximum concentration and baseline value for glycemia
Blood insulin peak | 4 hours
  Maximal concentration and delta between maximum concentration and baseline value for insulinemia

CONTACTS AND LOCATIONS:
Overall Officials: Jennie Brand Miller, Principal Investigator — University of Sydney
Locations (1):
- Human Nutrition Unit, The University of Sydney, Sydney, Australia